CLINICAL TRIAL: NCT04685733
Title: Caretaker Hemodynamic Parameters Validation
Status: Completed | Type: Observational
Sponsor: CareTaker Medical LLC (Industry)
Collaborators: University of Virginia (Other); Yale University (Other); Orange County Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: Hemo_001
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Blood Pressure; Cardiac Output; Left Ventricular Ejection Time; Heart Rate Variability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Group 1: Comparison of blood pressure, LVET and CO/SV measures with respective Gold Standards
  Interventions: Device: Non-invasive hemodynamic measurements
- Group 2: Comparison of blood pressure and HRV measures with respective Gold Standards
  Interventions: Device: Non-invasive hemodynamic measurements
- Group 3: Comparison of blood pressure and CO/SV measures with respective Gold Standards
  Interventions: Device: Non-invasive hemodynamic measurements

INTERVENTIONS:
Device: Non-invasive hemodynamic measurements — Non-invasive hemodynamic measurements

SUMMARY:
Comparison studies comparing hemodynamic parameters provided by the Caretaker against respective Gold Standard references.

DETAILED DESCRIPTION:
Comparison studies comparing hemodynamic parameters provided by the Caretaker against respective Gold Standard references.

Specifically, continuous beat-by-beat blood pressure readings against arterial catheter readings, continuous beat-by-beat left ventricular ejection times (LVET) against matching LVETs obtained from central catheters, cardiac output (CO) and stroke volume (SV) measures against thermo-dilution and Fick measurements, and standard HRV parameters based on Caretaker-provided inter-beat intervals (IBI) against the same HRV parameters obtained from ECG-based IBIs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age, who are able and willing to participate and have given written assent

Exclusion Criteria:

* Unable to give written assent

  * <18 years of age
  * No or poor finger pulse, as determined through visual inspection for ischemic hands

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be patients, > 18 years of age, who are able and willing to participate and have given written assent
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Blood pressure performance comparison | Paired beat-by-beat readings over maximum of 2.5 hours session length
  Comparison with arterial catheter-derived blood pressure, guidelines call for meeting a bias of 5 mmHg and a standard deviation of 8 mmHg
Cardiac output performance comparison | Paired measurements over approximately 1 hour time frame
  Comparison with thermo-dilution-based cardiac output, agreement within 1 l/min.
Left ventricular ejection time comparison | Paired measurements over approximately 1 hour time frame
  Comparison with LVET derived from central catheter signal traces, agreement within 20 msec.
Heart rate variability measures comparison | Paired beat-by-beat readings over maximum of 2.5 hours session length
  Comparison with 5 HRV ECG-derived measures, agreement within performance of VitalConnect predicate device

CONTACTS AND LOCATIONS:
Overall Officials: Martin Baruch, PhD, Principal Investigator — Caretaker Medical
Locations (1):
- Caretaker Medical, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided